CLINICAL TRIAL: NCT05427695
Title: Topical Probiotic Sinus Irrigations for the Treatment of Chronic Rhinosinusitis: a Double Blinded Randomized Controlled Trial
Brief Title: Topical Probiotic Sinus Irrigations for Treating Chronic Sinusitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, Victoria S. Lee, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-1205
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Adult patients of the PI's or co-investigator's with a diagnosis of active CRS and who meet the inclusion and exclusion criteria will be eligible to participate. A total of 60 subjects will be randomize evenly into 2 study groups: 30 patients in the saline group (SAL) and 30 patient in the Lactobacillus sakei group (LAC). Patients will asked to do nasal irrigations 2 times/day for 14 days. Patient history, sinus exams, culture swabs, surveys (SNOT-22) and pain scale will access pre and post treatment results. Patients will be assessed and compared prior to beginning sinus irrigations, the week after irrigations are completed, and 6 weeks after initial assessment.
Who Masked: Participant, Investigator
Masking Description: At the beginning of the study patients will be provided enough study product to complete 2 nasal sinus irrigations/day for a period of 14 days. There will be 1 packet for each nasal irrigation procedure (a total of 28 vials for 2 weeks). The packets will be distributed by the University's Investigational Drug Service (IDS) and will be labeled in a way that neither the patient nor the investigator will know the contents of the packet. Only IDS personnel will have the product/patient code link.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline Nasal Irrigation (Control) (Active Comparator): Patients will perform nasal irrigation with an isotonic saline solution, using a 240ml NeilMed sinus rinse bottle, 2 times/day for 14 days. A blinded packet supplied by IDS containing a premeasured amount of saline to be mixed with 240ml of distilled water will be provided to patients for each irrigation.
  Interventions: Other: Isotonic Saline Solution
- Lactobacillus sakei nasal irrigation (Experimental): Patients will perform nasal irrigation with Lactobacillus sakei, using a 240ml NeilMed sinus rinse bottle, 2 times/day for 14 days. A blinded packet provided by IDS containing a premeasured amount of Lactobacillus sakei to be mixed with 240ml of distilled water will be provided to patients for each irrigation.
  Interventions: Drug: Lactobacillus sakei proBio65

INTERVENTIONS:
Drug: Lactobacillus sakei proBio65 — Lanto Sinus probiotic Lactobacillus sakei is a currently available over the counter supplement from the common source kimchi and produced in South Korea. Patients will be instructed to mix 1 packet with lukewarm distilled or boiled water in 240mL NeilMed® sinus rinse bottle.
  Other Names: Lanto Sinus Probiotic Powder
  Arms: Lactobacillus sakei nasal irrigation
Other: Isotonic Saline Solution — Saline sinus irrigations (SAL group): NeilMed® Isotonic Sinus Rinse™ is marketed as a saline sinus irrigation formula. Subjects will be given instructions to mix one unlabeled packet (containing NeilMed® premixed buffered salt powder) with lukewarm distilled or boiled water in 240mL NeilMed® sinus rinse bottle.
  Other Names: NeilMed Isotonic Sinus Rinse
  Arms: Saline Nasal Irrigation (Control)

SUMMARY:
The purpose of this randomized study will be to determine whether topical probiotic sinus irrigations are more effective compared to saline sinus irrigation controls in the treatment of active CRS in patients who have had prior sinus surgery based on subjective and objective outcome measures.

DETAILED DESCRIPTION:
CRS is a common clinical entity with estimated prevalence ranging from 14-16% in the community. The most commonly implicated pathogenic bacteria in recalcitrant patients are Staphylococcus aureus (S. aureus) and Pseudomonas aeruginosa (P. aeruginosa). In recent years, there has been an increasing focus on the commensal sinonasal microbiome and its role in the development of a functional immune system. It has been theorized that infections in CRS may be related to a decrease in diversity of the commensal microbiome and an increase in these pathogenic bacteria. The concept behind the therapeutic potential of topical probiotics is that they outcompete pathogenic bacteria via a variety of mechanisms, including creating suboptimal environmental conditions, competing for cell surface receptors and thus limiting pathogen adherence, and producing antibacterial metabolites. In doing so, topical probiotics restore the commensal microbiome.

For this study, after being informed about the study and potential risks, all patients meeting eligibility criteria and giving written informed consent will be randomized in a double blind manner (participant and investigator) in a 1:1 ratio to Lactobacillus sakei or saline nasal irrigation, twice a day for 14 days.

Patient assessments will occur before treatments begin, immediately after the completion of nasal irrigations, and 6 weeks after initial enrollment. Assessments will be based on patient history, endoscopic exams, culture swab of the sinuses (bacterial burden and number of taxa, SNOT-22 survey, and a visual analog scale to record pain scores.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years of age or older.
2. Patients diagnosed with acute exacerbation of CRS, defined by worsening of 1 or more sinonasal symptoms (nasal obstruction/congestion, nasal discharge, facial pain/pressure, reduced sense of smell) and inflammatory and/or infectious changes on sinus endoscopy.
3. Patients that have undergone functional endoscopic sinus surgery > 12 months prior to enrollment as documented in the patients electronic medical record, with patent sinuses deemed suitable for trial on investigator's discretion.
4. Patients must be willing to follow study related procedures for the duration of the study.
5. Patients must understand the purpose and procedures and be willing to sign the study informed consent document.
6. All adult men and women with active CRS will be considered for participation in this study without regard to race, gender, or socioeconomic status.

Exclusion Criteria:

1. Patients who are taking topical antibiotic irrigations and are unwilling to stop them.
2. Patients who are unable to complete self-administered questionnaires because of cognitive impairment, language barrier, or severe medical conditions.
3. Patients who have a terminal illness (malignancy), immunocompromised (medication-related immunosuppression, immunodeficiency disorder) or systemic disease (granulomatosis polyangiitis or other autoimmune disease with sinonasal manifestations, cystic fibrosis), or recent head/sinonasal trauma that may predispose to infectious complications.
4. Patients who have severe or emergent complications from CRS or presence of a sinus tumor.
5. Female patients who are pregnant or breastfeeding. The patient will be asked if she is pregnant or has any chance of being pregnant. In either case, the patient will be excluded. Note in our consent form this is also addressed (excerpt below).
6. Patients who are taking oral corticosteroids or who have taken oral antibiotics in the previous 2 weeks or on oral corticosteroids.
7. Patients who have upper respiratory infection-type symptoms at time of enrollment, e.g., fevers/chills, sneezing, runny nose, sore throat, coughing. Patients can be eligible for enrollment once symptoms have fully resolved if all other inclusion/exclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Sinonasal Outcome Test-22 (SNOT-22) | 6 weeks
  It is expected that topical probiotic irrigations will result in a clinically significant change in symptom severity score (SNOT-22) (a change of 9 on a scale 0-110) compared to saline irrigations (primary outcome).

SECONDARY OUTCOMES:
Sinus microbiota | 6 weeks
  Nasal swab samples will be assessed for the number of bacteria present before and after treatment. Bacterial DNA will be extracted from nasal swabs. The purified DNA will be quantified for concentration using a Qubit fluorometer (Invitrogen, CA, USA) before storing at -20°C until further use. Bacterial burden will be determined by quantitative PCR (qPCR) using universal 16S ribosomal RNA primers. Additionally, each nasal swab will be assessed for bacteria taxonomic distribution by NGS using the MiSeq NGS platform (Illumina) before and after treatment. MiSeq paired-end sequencing of the hypervariable V3-V4 regions of the 16S rRNA gene (primers 341F/785R) will be performed.

OTHER OUTCOMES:
Lund-Kennedy Score | 6 weeks
  It is expected that topical probiotic irrigations will result in lower scores than sinus irrigations based on the Lund-Kennedy (LK) Endoscopic Scoring System. The LK system is used to evaluate sinus polyps, edema, discharge scarring and crusting. Scores range from 0 to 20. Lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Lee, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospitals & Health Sciences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee VS, Humphreys IM, Purcell PL, Davis GE. Manuka honey sinus irrigation for the treatment of chronic rhinosinusitis: a randomized controlled trial. Int Forum Allergy Rhinol. 2017 Apr;7(4):365-372. doi: 10.1002/alr.21898. Epub 2016 Dec 9. PMID 27935259
- [Background] Ooi ML, Jothin A, Bennett C, Ooi EH, Vreugde S, Psaltis AJ, Wormald PJ. Manuka honey sinus irrigations in recalcitrant chronic rhinosinusitis: phase 1 randomized, single-blinded, placebo-controlled trial. Int Forum Allergy Rhinol. 2019 Dec;9(12):1470-1477. doi: 10.1002/alr.22423. Epub 2019 Aug 28. PMID 31461581
- [Background] Orlandi RR, Kingdom TT, Hwang PH, Smith TL, Alt JA, Baroody FM, Batra PS, Bernal-Sprekelsen M, Bhattacharyya N, Chandra RK, Chiu A, Citardi MJ, Cohen NA, DelGaudio J, Desrosiers M, Dhong HJ, Douglas R, Ferguson B, Fokkens WJ, Georgalas C, Goldberg A, Gosepath J, Hamilos DL, Han JK, Harvey R, Hellings P, Hopkins C, Jankowski R, Javer AR, Kern R, Kountakis S, Kowalski ML, Lane A, Lanza DC, Lebowitz R, Lee HM, Lin SY, Lund V, Luong A, Mann W, Marple BF, McMains KC, Metson R, Naclerio R, Nayak JV, Otori N, Palmer JN, Parikh SR, Passali D, Peters A, Piccirillo J, Poetker DM, Psaltis AJ, Ramadan HH, Ramakrishnan VR, Riechelmann H, Roh HJ, Rudmik L, Sacks R, Schlosser RJ, Senior BA, Sindwani R, Stankiewicz JA, Stewart M, Tan BK, Toskala E, Voegels R, Wang de Y, Weitzel EK, Wise S, Woodworth BA, Wormald PJ, Wright ED, Zhou B, Kennedy DW. International Consensus Statement on Allergy and Rhinology: Rhinosinusitis. Int Forum Allergy Rhinol. 2016 Feb;6 Suppl 1:S22-209. doi: 10.1002/alr.21695. PMID 26889651
- [Background] Cervin AU. The Potential for Topical Probiotic Treatment of Chronic Rhinosinusitis, a Personal Perspective. Front Cell Infect Microbiol. 2018 Jan 12;7:530. doi: 10.3389/fcimb.2017.00530. eCollection 2017. PMID 29379772
- [Background] Foreman A, Psaltis AJ, Tan LW, Wormald PJ. Characterization of bacterial and fungal biofilms in chronic rhinosinusitis. Am J Rhinol Allergy. 2009 Nov-Dec;23(6):556-61. doi: 10.2500/ajra.2009.23.3413. PMID 19958600
- [Background] Gasta MG, Gossard CM, Williamson CB, Dolan KE, Finley HJ, Burns CM, Parker EC, Pizano JM, Lipski EA. Probiotics and Disease: A Comprehensive Summary-Part 5, Respiratory Conditions of the Ears, Nose, and Throat. Integr Med (Encinitas). 2017 Jun;16(3):28-40. PMID 30881245
- [Background] Abreu NA, Nagalingam NA, Song Y, Roediger FC, Pletcher SD, Goldberg AN, Lynch SV. Sinus microbiome diversity depletion and Corynebacterium tuberculostearicum enrichment mediates rhinosinusitis. Sci Transl Med. 2012 Sep 12;4(151):151ra124. doi: 10.1126/scitranslmed.3003783. PMID 22972842
- [Background] Humphreys GJ, McBain AJ. Antagonistic effects of Streptococcus and Lactobacillus probiotics in pharyngeal biofilms. Lett Appl Microbiol. 2019 Apr;68(4):303-312. doi: 10.1111/lam.13133. Epub 2019 Mar 13. PMID 30776138
- [Background] Forestier C, Guelon D, Cluytens V, Gillart T, Sirot J, De Champs C. Oral probiotic and prevention of Pseudomonas aeruginosa infections: a randomized, double-blind, placebo-controlled pilot study in intensive care unit patients. Crit Care. 2008;12(3):R69. doi: 10.1186/cc6907. Epub 2008 May 20. PMID 18489775
- [Background] Roos K, Hakansson EG, Holm S. Effect of recolonisation with "interfering" alpha streptococci on recurrences of acute and secretory otitis media in children: randomised placebo controlled trial. BMJ. 2001 Jan 27;322(7280):210-2. doi: 10.1136/bmj.322.7280.210. PMID 11159619
- [Background] Roos K, Simark-Mattsson C, Grahn Hakansson E, Larsson L, Sandberg T, Ahren C. Can probiotic lactobacilli eradicate persistent carriage of meticillin-resistant Staphylococcus aureus? J Hosp Infect. 2011 May;78(1):77-8. doi: 10.1016/j.jhin.2011.01.010. Epub 2011 Mar 2. No abstract available. PMID 21371778
- [Background] Bomer K, Brichta A, Baroody F, Boonlayangoor S, Li X, Naclerio RM. A mouse model of acute bacterial rhinosinusitis. Arch Otolaryngol Head Neck Surg. 1998 Nov;124(11):1227-32. doi: 10.1001/archotol.124.11.1227. PMID 9821924
- [Background] Prince AA, Steiger JD, Khalid AN, Dogrhamji L, Reger C, Eau Claire S, Chiu AG, Kennedy DW, Palmer JN, Cohen NA. Prevalence of biofilm-forming bacteria in chronic rhinosinusitis. Am J Rhinol. 2008 May-Jun;22(3):239-45. doi: 10.2500/ajr.2008.22.3180. PMID 18588755
- [Background] Rosenfeld RM. Clinical practice guideline on adult sinusitis. Otolaryngol Head Neck Surg. 2007 Sep;137(3):365-77. doi: 10.1016/j.otohns.2007.07.021. PMID 17765760
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277